CLINICAL TRIAL: NCT00442468
Title: An Evaluation of the Prevalence of Airway Obstruction Consistent With Chronic Obstructive Pulmonary Disease (COPD) in Subjects With a History of Cigarette Smoking and Symptoms of Chronic Bronchitis in a Primary Care Setting
Brief Title: Airway Limitation Study: Study In Primary Care Centers Of Chronic Bronchitis In Long-Term Cigarette Smokers Of At Least 40 Years Of Age With Symptoms Of Cough And Shortness Of Breath
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC109043
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Chronic Bronchitis; Spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- All participants: This is a cross-sectional, non-interventional study. All enrolled subjects were asked to complete a questionnaire and pulmonary function test to assess the prevalence of airflow obstruction.
  Interventions: Other: Non-interventional study.

INTERVENTIONS:
Other: Non-interventional study. — This is a non-interventional (no drug treatment administered), prevalence (observational) study.

SUMMARY:
The study does not involve testing of a drug (no treatment intervention). The study will will use spirometry (breathing tests) in subjects of 40 years of age and older with a history of cigarette smoking with chronic bronchitis to check their disease status and whether or not they have COPD. Also, study subjects will be asked to complete a questionnaire (to answer a list of questions on paper).

ELIGIBILITY:
Inclusion Criteria:

- Male or female - ≥40 years of age - Current or previous cigarette smoker with a history of cigarette smoking of ≥10 pack/years - Self reported symptoms of chronic bronchitis where chronic bronchitis is defined as the presence of productive cough for at least 3 months in each of the successive 2 years - Completion of written informed consent prior to study participation - Subject must be able to read, comprehend, and record information in English.

Exclusion Criteria:

- Regular use (i.e., prescribed for use on a daily basis) of the following respiratory medications for the six months prior to the study visit: ipratropium, ipratropium/albuterol combinations, tiotropium, salmeterol, formoterol, inhaled corticosteroids, inhaled corticosteroid/long-acting beta-agonist combinations, theophyllines, oral beta-agonists. - Previous lung surgery, including, lung transplant, lung resection, lung volume reduction surgery, etc. - Current diagnosis of a significant lung condition other than chronic bronchitis, including, asthma, lung cancer, cystic fibrosis, pulmonary fibrosis, bronchiectasis, active tuberculosis, sarcoidosis, or alpha-1-antitrypsin deficiency. - Any medical or physical condition that would interfere with the adequate performance of spirometry. - Evaluation and/or treatment by a pulmonary specialist (e.g., pulmonologist or allergist) within 3 years of the study visit. - A spirometrically confirmed diagnosis of COPD. - Have, in the opinion of the investigator, evidence of current alcohol, illegal drug or solvent abuse. - Limited ability to provide a valid informed consent due to serious uncontrolled psychiatric disease, intellectual or cognitive deficiency, poor motivation or other relevant condition which in the opinion of the site principal investigator will interfere with the subject's participation in the study. - Pregnant females. - Participating investigator, sub-investigator, study coordinator, employee of the participating investigator or family members of the aforementioned site staffs.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female, ≥40 years of age, current or previous cigarette smokers with ≥10 pack-years of smoking history and self reported symptoms of chronic bronchitis where chronic bronchitis.
Sampling Method: Probability Sample
Enrollment: 1283 (Actual)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (46):
  - GSK Investigational Site, Highlands Ranch, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Gillespie, Illinois
  - GSK Investigational Site, Vernon Hills, Illinois
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Nixa, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Fremont, Nebraska
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Mooresville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Sylva, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Beachwood, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Yukon, Oklahoma
  - GSK Investigational Site, Clairton, Pennsylvania
  - GSK Investigational Site, Harleysville, Pennsylvania
  - GSK Investigational Site, Cumberland, Rhode Island
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Harleysville, Tennessee
  - GSK Investigational Site, Milan, Tennessee
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Gig Harbor, Washington
  - GSK Investigational Site, Tacoma, Washington

REFERENCES:
- [Background] Yawn B, Mannino D, Littlejohn T, Ruoff G, Emmett A, Raphiou I, Crater G. Prevalence of COPD among symptomatic patients in a primary care setting. Curr Med Res Opin. 2009 Nov;25(11):2671-7. doi: 10.1185/03007990903241350. PMID 19757984

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants, With Self-reported Symptoms of Bronchitis: Participants with a minimum of 10 pack/year history of cigarette smoking and self-reported symptoms of chronic bronchitis in a primary care setting
Period: Overall Study
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Started | 1283
Completed | 1100
Not Completed | 183
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 91
Not completed — Did not complete all study procedures | 88

BASELINE CHARACTERISTICS:
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1283
Age Continuous [Mean (Standard Deviation); unit: years] | 52.9 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 704
  Male | 579
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European | 1030
  African American/African | 219
  White - Arabic/North African Heritage | 14
  American Indian or Alaskan Native | 13
  Mixed Race | 3
  Asian - Japanese | 2
  Asian - Central/South Central Asian Heritage | 1
  Native Hawain/Pacific Islander | 1
Smoking Status [Number; unit: participants] — Number of current and former smokers enrolled in the study
  participants
    Current smokers | 1116
    Former smokers | 167
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index (BMI, this is the ratio of the body mass in kilograms [kg] by the square of the height in meters [m2])
  kg/m2 | 28.7 (6.52)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Post-bronchodilator FEV1/FVC <=70% Versus Participants With a Postbronchodilator FEV1/FVC >70%
Description: Ratio of Forced Expiratory Volume in 1 second (volume of air expelled from the lungs in 1 second) by the Forced Vital Capacity (FVC, the volume of air that can forcibly be blown out after full inspiration) is a spirometric measure (lung function test) used to demonstrate airway obstruction. FEV1/FVC <=0.7 is used to demonstrate airway obstruction characteristic of chronic obstructive pulmonary disease (COPD).
Time Frame: Day 1 of a 1-day Study; before and 15-30 min after albuterol (self-administered under supervision of trained site staff)
Population: All enrolled participants who completed pre- and post-bronchodilator spirometry
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1201
participants
  FEV1/FVC<=70% | 308
  FEV1/FVC>70% | 893

2. Secondary Outcome: Number of Participants With the Indicated Scores on the MRC (Medical Research Council) Dyspnea Scale
Description: The MRC scale is a 6-point scale (scores from 0 to 5; encompassing degrees of dyspnea of none, slight, moderate, moderately severe, severe, and very severe) used to assess (via a participant-completed questionnaire) the amount of routine daily physical activity that precipitates dyspnea. The levels of physical activity range from strenuous exercise, to walking (including up a slight hill, on level ground, and to 100 yards), and to dressing and undressing.
Time Frame: Day 1 of a 1-day study
Population: All enrolled participants who completed the questionnaire
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1216
participants
  None (score=0) | 319
  Slight (score=1) | 572
  Moderate (score=2) | 254
  Moderately Severe (score=3) | 0
  Severe (score=4) | 68
  Very Severe (score=5) | 3

3. Secondary Outcome: Number of Participants With an Affirmative Response to Specific Categories on the Modified American Thoracic Society (ATS) Respiratory Questionnaire
Description: The Modified ATS Respiratory Questionnaire is a participant-completed questionnaire used to assess pulmonary disease symptomatology (such as cough, phlegm).
Time Frame: Day 1 of 1-day study
Population: All study participants who completed the questionnaire
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1283
participants
  Usually have cough | 1003
  Cough 4-6 times per day for at least 4 days/week | 917
  Cough when getting up first thing in the morning | 927
  Coughed during the rest of the day or night | 967
  Coughed most days for 3 consecutive months | 925
  Usually produced phlegm | 935
  Bring up phlegm twice/day for at least 4 days/week | 711
  Bring up phlegm first thing in the morning | 839
  Bring up phlegm during rest of the day or night | 718
  Bring up phlegm most days for 3 months | 764
  Had cough/phlegm episode for 3 or more weeks/year | 641
  Wheezy/whistling sound emanating from chest | 955
  Chest wheezing within week prior to study visit | 332
  Wheezing occuring with shortness of breath | 472
  Had a chest illness that kept them at home | 487
  Had a chest illness that produced phlegm | 656

4. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of How They'd Rate Their General Health, a Question on the 12-item Short Form Health Survey
Description: The 12-item short form health survey (SF-12, version 2) is a participant-completed questionnaire. The SF-12 Health Survey includes 12 questions from the SF-36 Health Survey. These include: 2 questions concerning physical functioning; 2 questions on role limitations because of physical health problems; 1 question on bodily pain; 1 question on general health perceptions; 1 question on vitality (energy/fatigue); 1 question on social functioning; 2 questions on role limitations because of emotional problems; and 2 questions on general mental health.
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1275
participants
  Excellent | 45
  Very good | 281
  Good | 675
  Fair | 236
  Poor | 38

5. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of Whether Their Health is Limited in Moderate Activities, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1272
participants
  Yes, limited a lot | 166
  Yes, limited a little | 437
  No, not limited at all | 669

6. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of Whether Their Health is Limited in Climbing Stairs, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1269
participants
  Yes, limited a lot | 336
  Yes, limited a little | 612
  No, not limited at all | 321

7. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of Whether They Had Accomplished Less Than They Would Like, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1276
participants
  All the time | 69
  Most of the time | 178
  Some of the time | 345
  A little of the time | 311
  None of the time | 373

8. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of How Often They Were Limited in the Kind of Work/Activities, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1272
participants
  All of the time | 91
  Most of the time | 144
  Some of the time | 334
  A little of the time | 264
  None of the time | 439

9. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of How Often They Accomplished Less Due to Emotional Problems, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1275
participants
  All of the time | 36
  Most of the time | 129
  Some of the time | 287
  A little of the time | 306
  None of the time | 517

10. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of How Often They Did Work Less Carefully Due to Emotional Problems, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1273
participants
  All of the time | 22
  Most of the time | 89
  Some of the time | 249
  A little of the time | 293
  None of the time | 620

11. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of to What Degree Does Pain Interfere With Normal Work, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1273
participants
  Not at all | 387
  A little bit | 258
  Moderately | 249
  Quite a bit | 207
  Extremely | 73

12. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of How Often They Felt Calm and Peaceful, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1273
participants
  All of the time | 84
  Most of the time | 595
  Some of the time | 372
  A little of the time | 172
  None of the time | 50

13. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of How Often They Have a Lot of Energy, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1265
participants
  All of the time | 58
  Most of the time | 367
  Some of the time | 446
  A little of the time | 300
  None of the time | 94

14. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of How Often They Felt Downhearted and Depressed, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1268
participants
  All of the time | 32
  Most of the time | 111
  Some of the time | 365
  A little of the time | 400
  None of the time | 357

15. Secondary Outcome: Number of Participants With the Indicated Responses to the Question of How Often They Experience Interference With Social Activities, a Question on the 12-item Short Form Health Survey
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the question
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1268
participants
  All of the time | 40
  Most of the time | 107
  Some of the time | 286
  A little of the time | 282
  None of the time | 553

16. Secondary Outcome: FEV1 and FVC, Pre-bronchodilator Spirometry Measures
Description: Participants self-administered a bronchodilator (albuterol) in the presence of trained site staff 15 to 30 minutes prior to pulmonary function test. FEV1 is the volume of air expelled from the lungs in 1 second, and FVC is the volume of air that can forcibly be blown out after full inspiration).
Time Frame: Day 1 of a 1-day study
Population: All participants who completed pre-bronchodilator spirometry
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1273
Liters (L)
  FEV1 | 2.46 (0.72)
  FVC | 3.46 (0.92)

17. Secondary Outcome: FEV1 Percent Predicted and FEV1/FVC Percent Predicted, Pre-bronchodilator Spirometry Measures
Description: Participants self-administered a bronchodilator (albuterol) in the presence of trained site staff 15 to 30 minutes prior to pulmonary function test. The FEV1 percent predicted and FEV1/FVC percent predicted are the test results as a percentage of the "predicted values" for participants of similar characteristics (height, age, sex, and sometimes race and weight).
Time Frame: Day 1 of a 1-day study
Population: All participants who completed pre-bronchodilator spirometry
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1273
percentage
  FEV1 percent predicted | 78.9 (17.21)
  FEV1/FVC percent predicted | 72.2 (8.77)

18. Secondary Outcome: FEV1 and FVC, Post-bronchodilator Spirometry Measures
Description: Participants completed the pulmonary function test 15-30 minutes after bronchodilator administration. FEV1 is the volume of air expelled from the lungs in 1 second, and FVC is the volume of air that can forcibly be blown out after full inspiration).
Time Frame: Day 1 of a 1-day visit
Population: All participants who completed post-bronchodilator spirometry
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1201
Liters
  FEV1 | 2.53 (0.73)
  FVC | 3.42 (0.91)

19. Secondary Outcome: FEV1 Percent Predicted and FEV1/FVC Percent Predicted, Post-bronchodilator Spirometry Measures
Description: Participants completed the pulmonary function test 15-30 minutes after bronchodilator administration. The FEV1 percent predicted and FEV1/FVC percent predicted are the test results as a percentage of the "predicted values" for participants of similar characteristics (height, age, sex, and sometimes race and weight).
Time Frame: Day 1 of a 1-day study
Population: All participants who completed pre- and post-bronchodilator spirometry
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1201
percentage
  FEV1 percent predicted | 81.4 (17.06)
  FEV1/FVC percent predicted | 74.0 (9.13)

20. Secondary Outcome: Post-bronchodilator Reversibility Measures
Description: To assess the reversibility in COPD, a bronchodilator was administered before performing another round of tests for comparison. This is commonly referred to as a reversibility test for the likelihood for a participant to revert to their baseline spirometric values or a post-bronchodilator test (Post BD) and is an important part in diagnosing asthma versus COPD, particularly since reversibility is not observed in the latter case. This differentiates COPD from other diseases.
Time Frame: Day 1 of a 1-day study
Population: All participants who completed pre- and post-bronchodilator spirometry
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1201
participants
  Non-reversible | 1088
  Reversible | 113

21. Secondary Outcome: Number of Participants Who Responded "Yes" to Respective Questions Regarding Past Illness
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the questions
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1283
participants
  Had lung trouble before age 16 | 62
  Ever had attack of bronchitis | 627
  Had an attack of bronchitis confirmed by doctor | 572
  Ever had sinus trouble | 743
  Had sinus trouble confirmed by doctor | 557
  Ever had tuberculosis | 11
  Had tuberculosis confirmed by doctor | 13
  Ever had pneumonia | 436
  Had pneumonia confirmed by doctor | 407
  Ever had fever | 274
  Had fever confirmed by doctor | 168
  Ever had asthma | 98
  Still have asthma | 40
  Had asthma confirmed by doctor | 88
  Ever hospitalized overnight for asthma | 15
  Hospitalized overnight for asthma in the last year | 4
  Ever had any other chest illness | 99
  Ever had any chest operation | 30
  Ever had any chest injury | 76
  Hospitalized for lung problems in past 12 months | 12
  Ever been treated with antibiotics for chest | 235

22. Secondary Outcome: Number of Participants Who Responded "Yes" to Respective Questions Regarding Occupational History and Socioeconomic Status
Time Frame: Day 1 of a 1-day study
Population: All participant respondents to the questions
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1283
participants
  Ever worked fulltime for more than 6 months | 1204
  Ever worked more than 1 year in any dusty job | 1246
  Ever been exposed to gas or chemical fumes | 433

23. Secondary Outcome: Number of Participants Who Completed the Highest Indicated Education Level or Grade
Time Frame: Day 1 of 1-day study
Population: All participant respondents to the questions
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1215
participants
  No or incomplete primary school | 5
  Completed primary school | 28
  Some high school | 163
  Completed high school | 468
  Technical post-secondary/further education | 358
  University graduate | 154
  University post-graduate degree | 39

24. Secondary Outcome: Number of Participants With the Indicated Experience With Tobacco Smoking
Time Frame: Day 1 of 1-day study
Population: All participant respondents to the questions
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1283
participants
  Ever smoked cigarettes | 1273
  Smoked cigarettes a month before study | 1092
  Smoked cigarettes in previous 24 hours | 1072
  Mother was a cigarette smoker | 761
  Father was a cigarette smoker | 949
  Smoked pipe regularly | 66
  Exposed to tobacco smoke from others | 788
  Anyone else smokes regularly at home | 583
  Anyone else smoked in childhood home | 1002

25. Secondary Outcome: Number of Participants Who Responded "Yes" When Asked Indicated Questions Regarding Medical History
Description: IBD, inflammatory bowel disease; GERD, gastroesophageal reflux disease.
Time Frame: Day 1 of 1-day study
Population: All participant respondents to the questions
Measure: Number; unit: participants
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Number analyzed (Participants) | 1283
participants
  Ever been told by a doctor you had heart trouble | 163
  Had treatment for heart trouble in past 10 years | 122
  Ever been told by doctor you had hypertension | 518
  Had treatment for hypertension in past 10 years | 434
  Ever been told by a doctor you had angina | 79
  Ever been told by a doctor you had a heart attack | 58
  Ever been told by a doctor you had a stroke | 31
  Ever been told by a doctor you had heart failure | 17
  Even been told by a doctor you had arrhythmia | 56
  Ever been told by a doctor you had osteoporosis | 96
  Ever been told by a doctor you had osteoarthritis | 190
  Ever been told by a doctor you had rheum arthritis | 119
  Ever been told by a doctor you had IBD | 76
  Ever been told by a doctor you had diabetes | 154
  Ever been told by a doctor you had Type I diabetes | 19
  Ever been told by doctor you had Type II diabetes | 124
  Ever been told by a doctor you had peptic ulcer | 70
  Ever been told by a doctor you had GERD | 45
  Ever had depression requiring treatment | 365
  Ever had anxiety/panic attacks | 325

ADVERSE EVENTS:
Time Frame: This is a single visit, non-interventional study; hence, AEs were collected during the visit.
Arm/Group | All Participants, With Self-reported Symptoms of Bronchitis
Serious Adverse Events (participants affected / at risk) | 0/1283
Other Adverse Events (participants affected / at risk) | 18/1283
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants, With Self-reported Symptoms of Bronchitis (N=1283)
Dizziness (Nervous system disorders) | 18
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.